CLINICAL TRIAL: NCT00939432
Title: The Greatest Taboo- Urinary Incontinence, Depression and Cancer
Brief Title: Taboo Perception of Incontinence, Depression and Cancer
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Engelbert Hanzal, MD Assoc Prof, Department of Obstetrics and Gynecology, Medical University of Vienna Austria
Other Study IDs: EK 453/2008
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Urinary Incontinence Awareness; Gender Differences
Keywords: incontinence; urinary; taboo; shame; embarrassment; treatment; depression; cancer
MeSH Terms: conditions — Depression; Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Gender: male/female
- Age: 18-100 years
- Educational level: primary school, secondary school, university

SUMMARY:
Objective/study hypothesis To evaluate how much of a taboo UI is and how it compares to other medical conditions that may also pose a taboo issue like depression and cancer.

Background Urinary incontinence (UI) is a highly prevalent condition with more than 200 million people worldwide being affected. While physical health does not necessarily have to be impaired much, restriction of social activities leads to isolation, a significant reduction in quality of life and will often bring about subsequent morbidity. Despite its prevalence, many patients suffering from UI go undiagnosed and untreated. Patients often hesitate to report the problem, and health care professionals often do not ask about it. In a study Minassian (2003) estimated that just one in four patients actively seeks medical attention. The reason for this may lie in the shame, embarrassment, and stigma associated with this condition, which in turn pose significant barriers to seeking professional treatment. Although mentioned by many narrative reviews and included in some epidemiological papers on UI, surprisingly we found no data addressing the taboo of UI exclusively. The aim of our study therefore was

Methods/Design A 13-question self-administered questionnaire was developed and face validity tested by 2 of the authors (KH, EH). The anonymous questionnaire contained simple questions on gender and age and then asked yes/no questions on whether test persons knew people with UI, or suspected other people to be incontinent, if they would address this issue with the suspected person, and if they thought that UI was a taboo issue in the society. On a scale from 0 - 10 they were then asked to grade the amount of embarrassment and anxiety if they themselves were incontinent, compared to depression or cancer. A few questions on knowledge of the condition of UI and to whom test persons would turn to in case of UI concluded the short questionnaire, which took about 5 minutes to fill in. A convenience sample of 150 test persons from waiting areas of a teaching hospital and in private practices of general practitioners in Austria agreed to take part in the study, with an additional 10 persons (6.2%) declining after being informed about the subject. Data were analysed with the SPSS 10.0.5 software package using the U-test, Chi-square-test, Yates-correction, Fisher's exact test and Kolmogorov-Smirnov normality test where appropriate.

ELIGIBILITY:
Inclusion Criteria:

- Subjects older than 18 years willing to take part in study mentally capable to understand and fill in anonymous questionnaire

Exclusion Criteria:

- incomplete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of 150 test persons from waiting areas of a teaching hospital and in private practices of general practitioners in Austria agreed to take part in the study, with an additional 10 persons (6.2%) declining after being informed about the subject.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-11; Primary Completion 2006-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Perception of given medical condition as a taboo issue | single point in time

SECONDARY OUTCOMES:
Knowledge of treatment options of incontinence | single point in time
Knowledge of friends or relatives with incontinence | single point in time

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna Austria, Vienna, Vienna, Austria